CLINICAL TRIAL: NCT03496688
Title: Comparative Histological and Histomorphometric Results of Six Biomaterials Used in Two-stage Maxillary Sinus Augmentation Model After 6-month-healing
Brief Title: Comparative Results of Six Biomaterials Used in Two-stage Maxillary Sinus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Maria Paola Cristalli, DDS PhD, Clinical Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3447/18.12.2014
Record Dates: First submitted 2018-03-29; First posted 2018-04-12 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Atrophy; Jaw, Edentulous, Partially; Sinus Floor Augmentation; Bone Substitutes; Bone Regeneration
Keywords: Sinus floor augmentation; Bone regeneration; Histology; Biocompatible materials; Bone transplantation
MeSH Terms: conditions — Atrophy; Jaw, Edentulous, Partially | interventions — Sinus Floor Augmentation

STUDY DESIGN:
Intervention Model Description: A randomized,controlled, double-blind clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant, Investigator, Outcome Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- bone substitute material MCBA (Active Comparator): Sinus floor augmentation: a bony window was created along the lateral wall of the sinus, the sinus membrane was carefully elevated and the created space was augmented using mineralized sol-vent-dehydrated bone allograft material.
  Interventions: Procedure: Sinus floor augmentation
- bone substitute material FDBA (Active Comparator): Sinus floor augmentation: a bony window was created along the lateral wall of the sinus, the sinus membrane was carefully elevated and the created space was augmented using freeze-dried mineralized bone allograft material.
  Interventions: Procedure: Sinus floor augmentation
- bone substitute material ABB (Active Comparator): Sinus floor augmentation: a bony window was created along the lateral wall of the sinus, the sinus membrane was carefully elevated and the created space was augmented using anorganic bovine bone material.
  Interventions: Procedure: Sinus floor augmentation
- bone substitute material EB (Active Comparator): Sinus floor augmentation: a bony window was created along the lateral wall of the sinus, the sinus membrane was carefully elevated and the created space was augmented using equine-derived bone material.
  Interventions: Procedure: Sinus floor augmentation
- bone substitute material HA-β-TCP 30/70 (Active Comparator): Sinus floor augmentation: a bony window was created along the lateral wall of the sinus, the sinus membrane was carefully elevated and the created space was augmented using synthetic micromacroporous bi-phasic calcium-phosphate block consisting of 70% beta-tricalcium phosphate and 30% hy-droxyapatite material.
  Interventions: Procedure: Sinus floor augmentation
- bone substitute material BC (Active Comparator): Sinus floor augmentation: a bony window was created along the lateral wall of the sinus, the sinus membrane was carefully elevated and the created space was augmented using bioapatite-collagen material.
  Interventions: Procedure: Sinus floor augmentation

INTERVENTIONS:
Procedure: Sinus floor augmentation

SUMMARY:
Objectives: The aim of the study was to compare histological and histomorphometric results of six bone substitute materials used as graft in two-stage maxillary sinus augmentation model, after 6-month-healing.

DETAILED DESCRIPTION:
Materials and Methods:

A two-stage sinus augmentation was carried out in six patients using mineralized solvent-dehydrated bone allograft (MCBA), freeze-dried mineralized bone allograft (FDBA), anor-ganic bovine bone (ABB), equine-derived bone (EB); synthetic micromacroporous biphasic calcium-phosphate block consisting of 70% beta-tricalcium phosphate and 30% hydroxyap-atite (HA-β-TCP 30/70), or bioapatite-collagen (BC).

ELIGIBILITY:
Inclusion Criteria: patients healthy, absence of systemic pathologies (ASA class I), non-smokers, good oral hygiene, not pregnant or lactating, absence of painful symptoms and associated inflammatory or osteolytic pathologies, maxillary partial edentulism involving the premolar/molar areas, residual bone height between the sinus floor and alveolar ridge ranging from 2 to 4 mm, as measured on computerized tomography (CT) scan.

-

Exclusion Criteria:

-

Ages: 33 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2016-01-04 (Actual); Study Completion 2017-09-11 (Actual)

PRIMARY OUTCOMES:
to perform biopsies from each six augmented site using to compare, histologically and histomorphometrically, the percentages of newly formed bone, residual grafted material, and marrow spaces. | 6 month-healing after surgery
  After 6 months clinical and radiographic examinations were undertaken and each patient was reappointed for biopsy at the time of implant placement in the same location. Under local anesthesia, a full thickness flap was raised, a biopsy was performed using a 3.5 mm tre-phine bur under sterile saline solution irrigation, guided by the radiographic/surgical template in the selected implant site. A total of six bone samples was retrieved from the occlusal aspect to the alveolar crest, one from each augmented site to compare histologically and histomorphometrically the different materials.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Paola Cristalli, DDS, Principal Investigator — University of Roma La Sapienza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] La Monaca G, Iezzi G, Cristalli MP, Pranno N, Sfasciotti GL, Vozza I. Comparative Histological and Histomorphometric Results of Six Biomaterials Used in Two-Stage Maxillary Sinus Augmentation Model after 6-Month Healing. Biomed Res Int. 2018 Jun 27;2018:9430989. doi: 10.1155/2018/9430989. eCollection 2018. PMID 30050947